CLINICAL TRIAL: NCT04597684
Title: What Are the Results of Cemented vs. Cementless TKA With the Same Implant Design? A Randomized Clinical Trial.
Brief Title: Cemented vs. Cementless TKA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment volume below acceptable accrual rate.
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HK226
Record Dates: First submitted 2020-10-09; First posted 2020-10-22 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Total Knee Arthroplasty (TKA)
MeSH Terms: interventions — Therapeutics; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment/Intervention (Active Comparator): Total Knee Arthroplasty (TKA) with cementless knees
  Interventions: Procedure: Cementless Total Knee Arthroplasty
- Control (Active Comparator): Total Knee Arthroplasty (TKA) with cemented knees
  Interventions: Procedure: Cemented Total Knee Arthroplasty

INTERVENTIONS:
Procedure: Cementless Total Knee Arthroplasty — Total Knee Arthroplasty (TKA) with cementless knees
  Other Names: Treatment/Intervention
  Arms: Treatment/Intervention
Procedure: Cemented Total Knee Arthroplasty — Total Knee Arthroplasty (TKA) with cemented knees
  Other Names: Control
  Arms: Control

SUMMARY:
The investigators are evaluating an implant (Depuy Attune TKA) that was recently released to market with a cementless design that is yet to have long term comparative data between this cementless design or cemented options. The investigators are conducting a study to compare the results of this cementless design to the cemented design of the same implant.

DETAILED DESCRIPTION:
Aseptic Loosening remains a leading cause for revision following TKA. Cemented TKAs have shown high failure rates in obese and younger populations. There is renewed interest in biologic fixation of total knee components with a more active and younger patient population, as well as long term alternatives in obese patients receiving TKA.

Questions remain whether cemented or cementless long term fixation is superior in total knee arthroplasty in these populations.

Potential benefits of cementless fixation include preservation of bone, decreased operative times, and elimination of complications specific to cemented components. Older cementless TKA designs had higher failure rates due to poor fixation methods, patch porous coating on the implant, poor tibial locking mechanisms and the use of conventional polyethylene. The combination of these factors led to unacceptable failure rates in these devices. Newer designs have looked to improve these flaws with advances in the biologic interface, use of highly porous metals, improved locking mechanisms, and cross-linked polyethylene.

Recently, cementless implants with these improved design features have shown improved long term outcomes of cementless components versus their cemented predecessors. The combination of these improved long term outcomes in younger, more active population warrant further investigation of cementless components in TKA. There is a need for more durable, long term fixation in all implants treating obese, as well as young active patients.

The investigators are evaluating an implant (Depuy Attune TKA) that was recently released to market with a cementless design that is yet to have long term comparative data between this cementless design or cemented options. The investigators are conducting a study to compare the results of this cementless design to the cemented design of the same implant.

ELIGIBILITY:
Inclusion Criteria:

1. Evaluation for TKA at OrthoCarolina
2. Evaluated and scheduled for TKA by Drs. Keith Fehring, Bo Mason, William Griffin, Thomas Fehring, or Jesse Otero
3. Determined by the above surgeon to be a candidate for the Attune Posterior Stabilized knee system, with the patella to be resurfaced during surgery
4. >18 years of age at enrollment

Exclusion Criteria:

1. Previous surgery with hardware on the joint of interest
2. >= 65 years old at the time of TKA surgery
3. Previous diagnosis of inflammatory disease (RA, inflammatory arthropathy, any autoimmune disease)
4. BMI <= 40
5. Physician discretion due to not being able to follow standard-of-care (SOC) TKA follow up protocol
6. History of contralateral TKA
7. Current Tobacco Use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Revision for loosening | Within 20 years of study surgery
  Did the subject have a revision procedure due to loosening (yes/no)

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS Jr.) | PreOperative, 3 months, 6 months, 1 year, 2 year, 5 year, 10 year, 15 year, 20 year
  Patient-reported outcome of knee stiffness, pain, and function of daily living.
The Veterans RAND 12-Item Health Survey (VR-12) | PreOperative, 3 months, 6 months, 1 year, 2 year, 5 year, 10 year, 15 year, 20 year
  General Health survey
Radiographic evidence of loosening | PreOperative, 3 months, 6 months, 1 year, 2 year, 5 year, 10 year, 15 year, 20 year
  Radiographic evidence of loosening

OTHER OUTCOMES:
Charlson Comorbidity Index (CCI) | PreOperative
  Evaluation of a subject's mortality risk

CONTACTS AND LOCATIONS:
Overall Officials: Keith A Fehring, MD, Principal Investigator — OrthoCarolina Research Institute, Inc.
Locations (1):
- OrthoCarolina Research Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared with other researchers.

REFERENCES:
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Miller AJ, Stimac JD, Smith LS, Feher AW, Yakkanti MR, Malkani AL. Results of Cemented vs Cementless Primary Total Knee Arthroplasty Using the Same Implant Design. J Arthroplasty. 2018 Apr;33(4):1089-1093. doi: 10.1016/j.arth.2017.11.048. Epub 2017 Dec 2. PMID 29275115
- [Background] Nam D, Lawrie CM, Salih R, Nahhas CR, Barrack RL, Nunley RM. Cemented Versus Cementless Total Knee Arthroplasty of the Same Modern Design: A Prospective, Randomized Trial. J Bone Joint Surg Am. 2019 Jul 3;101(13):1185-1192. doi: 10.2106/JBJS.18.01162. PMID 31274720
- [Background] Fricka KB, Sritulanondha S, McAsey CJ. To Cement or Not? Two-Year Results of a Prospective, Randomized Study Comparing Cemented Vs. Cementless Total Knee Arthroplasty (TKA). J Arthroplasty. 2015 Sep;30(9 Suppl):55-8. doi: 10.1016/j.arth.2015.04.049. Epub 2015 Jun 3. PMID 26118567
- [Background] Abdel MP, Bonadurer GF 3rd, Jennings MT, Hanssen AD. Increased Aseptic Tibial Failures in Patients With a BMI >/=35 and Well-Aligned Total Knee Arthroplasties. J Arthroplasty. 2015 Dec;30(12):2181-4. doi: 10.1016/j.arth.2015.06.057. Epub 2015 Jul 2. PMID 26220103
- [Background] Carr AJ, Robertsson O, Graves S, Price AJ, Arden NK, Judge A, Beard DJ. Knee replacement. Lancet. 2012 Apr 7;379(9823):1331-40. doi: 10.1016/S0140-6736(11)60752-6. Epub 2012 Mar 6. PMID 22398175
- [Background] Brown TE, Harper BL, Bjorgul K. Comparison of cemented and uncemented fixation in total knee arthroplasty. Orthopedics. 2013 May;36(5):380-7. doi: 10.3928/01477447-20130426-10. PMID 23672897
- [Background] Lombardi AV Jr, Berasi CC, Berend KR. Evolution of tibial fixation in total knee arthroplasty. J Arthroplasty. 2007 Jun;22(4 Suppl 1):25-9. doi: 10.1016/j.arth.2007.02.006. PMID 17570273